CLINICAL TRIAL: NCT03143972
Title: Pharmacodynamic Interactions Between Remifentanil and Dexmedetomidine (PIRAD)
Brief Title: Pharmacodynamic Interaction of REMI and DMED
Acronym: PIRAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PIRAD-001
Record Dates: First submitted 2017-03-14; First posted 2017-05-08 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia
Keywords: Dexmedetomidine; Remifentanil; Pharmacodynamics; Interaction
MeSH Terms: interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Intervention Model Description: All volunteers will receive 2 standardized anesthesia sessions with a washout period of at least one week between sessions. During the first session volunteers will receive dexmedetomidine, during the second session they will first receive remifentanil and afterwards the combination of drugs will be administered. Anesthetic depth will be evaluated by MOAA/S scores (see table 2), testing of tolerance to electrical stimuli and laryngoscopy. Furthermore multichannel EEG-data will be collected to get insight in the drug dependent characteristics. Measured effects will be related to drug plasma concentrations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine only (Experimental): Dexmedetomidine will be administered by effect-site TCI according to the Hannivoort model extended with an effect-site rate constant of 0.0428min-1.
  A stepwise increasing dosing regimen will be given, with concentrations targeting an effect site concentration of 1 ng/ml (40 min), 3 ng/ml (50 min), 4 ng/ml (40 min), 5 ng/ml (40 min) and 8 ng/ml (70 min).
  Interventions: Drug: Dexmedetomidine
- Remifentanil only (Experimental): Remifentanil will be administered by effect-site TCI according to the Eleveld model. A stepwise increasing dosing regimen will be given, with concentrations targeting an effect site concentration of 1 ng/ml (12 min), 2 ng/ml (12 min), 3 ng/ml (12 min), 5 ng/ml (12 min) and 7 ng/ml (12 min).
  Interventions: Drug: Remifentanil
- Dexmedetomidine-Remifentanil interaction (Experimental): A fixed background dose of dexmedetomidine will be given, this will be calculated after the first 5 subjects completed the dexmedetomidine only session. It will be set to 50% of the observed mean EC50TOL (Tolerance of Laryngoscopy).
  Remifentanil infusion will be administered by effect site TCI with stepwise increasing targets of 0.5 - 1.0 - 1.5 - 2.0 - 2.5 - 3.0 - 4.0 ng/ml, each lasting for 15 minutes.
  Interventions: Drug: Dexmedetomidine; Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — Single drug administration
  Other Names: Dexdor
  Arms: Dexmedetomidine only; Dexmedetomidine-Remifentanil interaction
Drug: Remifentanil — Single drug administration
  Other Names: Ultiva
  Arms: Dexmedetomidine-Remifentanil interaction; Remifentanil only

SUMMARY:
The objective is to map the pharmacokinetic / pharmacodynamic interaction between dexmedetomidine and remifentanil by observing changes in anesthetic depth. These changes will be related to drug concentrations using pharmacokinetic/pharmacodynamic (PKPD) modeling.

DETAILED DESCRIPTION:
This study is designed to investigate whether the use of a combination of dexmedetomidine and remifentanil is clinically useful to provide anesthesia during surgical and diagnostic procedures and whether it could be used for anesthetic induction. Furthermore the aim is to gain better insights in the required dosing regimens, the inter-individual variability in response towards the combination and the associated side effects. Better characterization of this drug-drug interaction will presumably lead to more precise dosing regimens, which in turn, will lead to a reduction in the occurrence of oversedation, side effects and recovery times.

The objective is to map the pharmacokinetic / pharmacodynamic interaction between dexmedetomidine and remifentanil by observing changes in anesthetic depth, measured by hypnotic and analgesic endpoints such as modified observer's assessment of alertness and sedation scale (MOAA/S), response to electrical stimuli, response to laryngoscopy and electroencephalogram (EEG) derived indices. These effects will be related to drug concentrations using pharmacokinetic/pharmacodynamic (PKPD) modeling.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status 1
* No medical history of significance
* No chronic use of medication, drugs, tobacco or more than 20 gr alcohol daily (oral contraceptives excluded).
* Concerning the cognitive function: Volunteers are considered to have sufficient cognitive reserve if they are able to read and comprehend the patient information form, if they can adequately answer the anamnestic questions during the screening process and if they are allowed to provide legitimate written informed consent.
* No selection will be made regarding ethnic background
* No exclusion criterium is present

Exclusion Criteria:

* Known intolerance to dexmedetomidine or remifentanil
* Volunteer refusal
* Age < 18 years or >70 years
* Pregnancy, or currently nursing
* Hairstyle with dreadlocks (EEG-monitoring will not be possible)
* Body mass index (BMI) <18 or >30 kg/m2.
* Neurological disorder (epilepsy, the presence of a brain tumor, a history of brain surgery, hydrocephalic disorders, depression needing treatment with anti-depressive drugs, a history of brain trauma, a subarachnoidal bleeding, TIA or cerebral infarct, psychosis or dementia , schizophrenia, alcohol or drug abuse).
* Diseases involving the cardiovascular system (hypertension, coronary artery disease, prior acute myocardial infarction, any valvular and/or myocardial disease involving

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Tolerance of Laryngoscopy (TOL) | 35 - 255 minutes
  Tolerance of a laryngoscopy (yes/no) will be tested at the end of each infusion step during both studydays, when MOAA/s is 0 / 1 and will be related to the drug concentration(s).

SECONDARY OUTCOMES:
Modified observer's assessment of alertness and sedation scale (MOAA/s) | During anesthesia sessions day 1 and day 2
  An hypnotic endpoint measuring depth of anesthesia.
Electrical stimulus | During anesthesia sessions day 1 and day 2
  Measuring analgesia by observing response to a standardized electrical stimulus
Electroencephalogram (EEG) | During anesthesia sessions day 1 and day 2
  A multichannel electroencephalogram will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Michel MR Struys, Prof.Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Anonimous data might be shared with other research groups

REFERENCES:
- [Background] Hannivoort LN, Eleveld DJ, Proost JH, Reyntjens KM, Absalom AR, Vereecke HE, Struys MM. Development of an Optimized Pharmacokinetic Model of Dexmedetomidine Using Target-controlled Infusion in Healthy Volunteers. Anesthesiology. 2015 Aug;123(2):357-67. doi: 10.1097/ALN.0000000000000740. PMID 26068206
- [Derived] Su H, Koomen JV, Eleveld DJ, Struys MMRF, Colin PJ. Pharmacodynamic mechanism-based interaction model for the haemodynamic effects of remifentanil and propofol in healthy volunteers. Br J Anaesth. 2023 Aug;131(2):222-233. doi: 10.1016/j.bja.2023.04.043. Epub 2023 Jun 22. PMID 37355412
- [Derived] Ramaswamy SM, Kuizenga MH, Weerink MAS, Vereecke HEM, Struys MMRF, Belur Nagaraj S. Frontal electroencephalogram based drug, sex, and age independent sedation level prediction using non-linear machine learning algorithms. J Clin Monit Comput. 2022 Feb;36(1):121-130. doi: 10.1007/s10877-020-00627-3. Epub 2020 Dec 14. PMID 33315176
- [Derived] Ramaswamy SM, Weerink MAS, Struys MMRF, Nagaraj SB. Dexmedetomidine-induced deep sedation mimics non-rapid eye movement stage 3 sleep: large-scale validation using machine learning. Sleep. 2021 Feb 12;44(2):zsaa167. doi: 10.1093/sleep/zsaa167. PMID 32860500
- [Derived] Belur Nagaraj S, Ramaswamy SM, Weerink MAS, Struys MMRF. Predicting Deep Hypnotic State From Sleep Brain Rhythms Using Deep Learning: A Data-Repurposing Approach. Anesth Analg. 2020 May;130(5):1211-1221. doi: 10.1213/ANE.0000000000004651. PMID 32287128
- [Derived] Ramaswamy SM, Kuizenga MH, Weerink MAS, Vereecke HEM, Struys MMRF, Nagaraj SB. Novel drug-independent sedation level estimation based on machine learning of quantitative frontal electroencephalogram features in healthy volunteers. Br J Anaesth. 2019 Oct;123(4):479-487. doi: 10.1016/j.bja.2019.06.004. Epub 2019 Jul 18. PMID 31326088